CLINICAL TRIAL: NCT01792882
Title: Prospective Collection of Surplus Surgical Tumor Tissues and Pre-surgical Blood Samples
Acronym: GBCPRT0008
Status: Withdrawn | Type: Observational
Sponsor: Global BioClinical (Industry)
Responsible Party: Sponsor
Other Study IDs: GBC PRT0008
Record Dates: First submitted 2013-02-06; First posted 2013-02-15 (Estimated); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer; Colorectal Cancer; Lung Cancer; Prostate Cancer; Hematologic Cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Lung Neoplasms; Prostatic Neoplasms; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Surplus Surgical Tissues
  Tissue procurement will involve the collection of tissues snap frozen in liquid nitrogen. Tissues will include tumors and histologically normal (uninvolved) areas (>2cm from tumor) of tissue. A tumor tissue sample is required; a normal tissue sample should be provided if available.
  Individual samples will be collected in weights (sizes) approximately 100-200 mg or larger. Research tissues sample collection will only be performed on surplus (discard) tissues not required for patient diagnosis and will never interfere with clinical diagnosis.
  Blood Samples
  Blood samples will be collected from consented subjects prior to surgery and will involve the collection of up to 20 ml of whole blood into appropriate blood collection tubes and freezing them.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cancer Subjects

SUMMARY:
The study is intended to collect specimens to support the application of genome analysis technologies, including large-scale genome sequencing. This study will ultimately provide cancer researchers with specimens that they can use to develop comprehensive catalogs of genomic information on at least 50 types of human cancer. The study will create a resource available to the worldwide research community that could be used to identify and accelerate the development of new diagnostic and prognostic markers, new targets for pharmaceutical interventions, and new cancer prevention and treatment strategies. This study will be a competitive enrollment study conducted at multiple institutions.

DETAILED DESCRIPTION:
This study will enroll subjects diagnosed with various cancers and who are scheduled to undergo surgical treatment. Prior to scheduled surgery, subjects will be asked to donate a 10-20 ml blood sample. After surgery, surplus tissues (including tumor and adjacent normal tissues) not required for diagnosis will be collected. Subject clinical information will be collected, including basic demographic information, medical history, family history, current cancer history and treatment. After surgery, a final pathology report will be obtained for each subject's surgical specimen. In some instances and based on the cancer indications required, longitudinal data may also be collected at a frequency of every 6 months to once per year. Longitudinal data will include information on study subject survival and disease recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Any adult age
* Any sex
* Able to provide consent for surplus tissue and/or blood donation
* Diagnosed with one of the cancer indications listed below:
* Scheduled to undergo surgical resection of tumor (exception for hematological cancers)
* Have not yet received treatment for cancer

Exclusion Criteria:

* Not diagnosed with required cancer indication
* Not scheduled to undergo surgical resection of the tumor
* Have already received cancer treatment (such as chemotherapy, radiation, surgery) for the current cancer or a previously diagnosed cancer
* Not able to donate an adequate volume of blood to meet minimum requirements

CANCER INDICATIONS:

1. Bladder Cancer - Urothelial carcinoma - nonpapillary
2. Bladder Cancer - Urothelial carcinoma - papillary
3. Brain Cancer - Astrocytoma
4. Brain Cancer - Glioblastoma
5. Brain Cancer - Medulloblastoma
6. Breast Cancer - Ductal Carcinoma
7. Breast Cancer - Lobular Carcinoma
8. Cervical Cancer - Squamous Cell Carcinoma
9. Colorectal Cancer - Adenocarcinoma
10. Esophageal Cancer - Adenocarcinoma
11. Gastric Cancer
12. Head and Neck Cancer - Squamous Cell Carcinoma
13. Hematologic Cancer - Acute Lymphocytic Leukemia (ALL)
14. Hematologic Cancer - Acute Myeloid Leukemia (AML)
15. Hematologic Cancer - Chronic Lymphocytic Leukemia (CLL)
16. Hematologic Cancer - Diffuse Large B-cell Lymphoma
17. Hematologic Cancer - Multiple Myeloma (MM)
18. Hematologic Cancer - Non-Hodgkins Lymphoma (NHL)
19. Kidney Cancer - Papillary Carcinoma
20. Kidney Cancer - Renal cell Carcinoma
21. Liver Cancer - Hepatocellular Carcinoma
22. Lung Cancer - Adenocarcinoma
23. Lung Cancer - Squamous Cell Cancer
24. Melanoma
25. Pancreatic Cancer - Ductal Adenocarcinoma
26. Prostate Cancer - Adenocarcinoma
27. Sarcomas
28. Thyroid Cancer - Follicular Carcinoma
29. Thyroid Cancer - Papillary Carcinoma
30. Uterine Cancer - Endometrial Carcinoma

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects diagnosed with one of the cancer indications listed below and scheduled to undergo surgical tumor resection
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-02; Primary Completion 2022-12-31 (Actual); Study Completion 2023-02-27 (Actual)

PRIMARY OUTCOMES:
Tumor genetic sequence variation | up to 18 months
  The specimens collected for this project will support genomic studies on the molecular basis of cancer. This study aims to collect specimens for a project that will systematically explore a spectrum of genomic changes involved in human cancer. Specifically the project will analyze DNA copy number changes, including large (on the order of chromosomal segments) and small (1,000 to 100,000 KB) scale rearrangements, transcription profiles, epigenetic modifications, sequence variation, and sequence in both tumor tissue and case-matched germline DNA. The suite of analysis platforms for collaborating laboratories will be applied to a common set of molecular analytes obtained from clinically annotated high-quality tumor specimens and case matched normal control specimens obtained form this specimen collection study. Initial measures critical to ensure specimen quality and qualification for subsequent analysis include confirmed histopathology and RNA integrity.

SECONDARY OUTCOMES:
Transcription profile | up to 18 months

OTHER OUTCOMES:
Epigenetic modification | up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Neil R Mucci, Study Director — Global BioClinical
Locations (1):
- GBC, Seattle, Washington, United States